CLINICAL TRIAL: NCT01519440
Title: Unintended Extension of the Lower Segment Uterine Incision at Cesarean Delivery;A Randomized Comparison of Sharp Versus Blunt Techniques
Brief Title: Randomized Comparison of Sharp Versus Blunt Techniques at Cesarean
Status: Completed | Type: Observational
Sponsor: Istanbul Bakirkoy Maternity and Children Diseases Hospital (Other Government)
Responsible Party: Principal Investigator, Osman Aşıcıoğlu, MD, Istanbul Bakirkoy Maternity and Children Diseases Hospital
Other Study IDs: Aşıcıoğlu-01
Record Dates: First submitted 2012-01-24; First posted 2012-01-27 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Disruption of Uterine Incision After Cesarean Section
Keywords: unintended extension; blunt; sharp; maternal blood loss

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

GROUPS / COHORTS (2):
- blunt: Blunt expansion of the primary incision was derived by placing the index fingers of the operating surgeon into the incision and pulling the fingers apart laterally and cephalad.
- sharp: Sharp expansion of the primary incision was developed by cutting laterally and cephalad using bandage scissors

SUMMARY:
The purpose of this study is to determine whether a specific surgical technique, blunt compared with sharp expansion of the transverse lower uterine incision, is associated with risk of unintended extension of uterine incision

ELIGIBILITY:
Inclusion Criteria:

1. Term pregnancy(> 38 weeks of gestation)
2. Required elective cesarean delivery
3. maternal age between 18-40 years

Exclusion Criteria:

1. Required emergency cesarean delivery
2. Abnormal presentation
3. Planned cesarean hysterectomy
4. History of low segment vertical uterine incision
5. History of classical upper segment uterine incision
6. multiple pregnancy
7. cases with a high risk for bleeding(HELLP send, preeclampsia, placental insertion anomalies)
8. Grand multiparity(parity>5)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: elective cesarean delivery cases
Sampling Method: Probability Sample
Enrollment: 1076 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
unintended extension of uterine incision | during the operation

SECONDARY OUTCOMES:
intraoperative maternal blood loss | after 48 hours than operation

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Bakırköy Maternal and Childrens Hospital, Istanbul, Bakırköy, Turkey (Türkiye)

REFERENCES:
- [Result] Magann EF, Chauhan SP, Bufkin L, Field K, Roberts WE, Martin JN Jr. Intra-operative haemorrhage by blunt versus sharp expansion of the uterine incision at caesarean delivery: a randomised clinical trial. BJOG. 2002 Apr;109(4):448-52. doi: 10.1111/j.1471-0528.2002.01296.x. PMID 12013167